CLINICAL TRIAL: NCT00270712
Title: Study of Long-term Deterioration of Kidney Allograft Function (DeKAF)
Brief Title: A Study of Factors That Affect Long-Term Kidney Transplant Function
Acronym: DeKAF
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Astellas Pharma Inc (Industry); Bristol-Myers Squibb (Industry); Novartis (Industry); Pfizer (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 0407M62262
Record Dates: First submitted 2005-12-27; First posted 2005-12-28 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Kidney Transplant
Keywords: kidney; transplant; dysfunction; chronic; deterioration; loss of function
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood and urine specimens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective Cohort: 537 transplant recipient records used retrospectively
- Prospective Cohort: 3137 transplant recipients enrolled prospectively

SUMMARY:
The causes of deterioration of transplanted kidney function are poorly understood. The purpose of this study is to determine the disease processes that cause transplanted kidney dysfunction and loss in patients who received a kidney either recently or over a year prior to entering this study. This study will also identify specific characteristics in kidney transplant recipients that predict whether a kidney transplant will be successful.

DETAILED DESCRIPTION:
Over time, chronic kidney graft dysfunction progressively threatens the long-term survival of a kidney graft. The disease processes behind graft dysfunction are unclear. However, chronic kidney graft dysfunction is likely to be caused by certain definable factors. Such factors may include collagens III and IV, transforming growth factor (TGF)-beta, T and B cell surface markers, cell cycle proteins, fibronectin, and laminin. Determining what disease processes and which specific factors are most responsible for kidney graft dysfunction may help in designing future interventional trials for kidney transplant patients. The purpose of this study is to determine whether clinical, laboratory, and histologic studies at the time of initial graft dysfunction will clarify the processes and factors that lead to deterioration and loss of a kidney graft. This is an observational study that will enroll participants who have recently received kidney transplants (prospective cohort) and participants who have had kidney transplants for a longer period of time and are now experiencing kidney graft dysfunction (retrospective cohort).

The duration of this trial may differ between participants, depending on when deterioration of kidney graft function occurs. Participants will be followed until graft loss or death. There are no exclusive study visits associated with this study. Study data are gathered from routine laboratory follow-up tests completed at the participant's local medical center and from information obtained at the time of kidney biopsy. Participants may need to undergo a kidney biopsy as clinically indicated. At the time of biopsy, participants will also undergo urine and blood collection.

ELIGIBILITY:
Inclusion Criteria for Prospective Cohort:

* Received a kidney transplant within 10 days prior to study entry, on or after 10-01-2005
* Recipient of kidney or simultaneous kidney/pancreas with no additional transplant at the time of the kidney transplant

Inclusion Criteria for Retrospective Cohort:

* Received a kidney transplant before 10-01-2005
* Recipient of kidney or simultaneous kidney/pancreas with no additional transplant at the time of the kidney transplant
* Undergoes a clinically indicated kidney biopsy due to new onset deterioration of function, defined as having an increase in serum creatinine
* The creatinine level on or before 01-01-2006 must be 2 mg/dl or less OR the patient must have developed new onset proteinuria, defined as having a protein/creatinine ratio of 0.4 or more

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 3175 (Actual)
Dates: Start 2005-10; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Kidney transplant failure | throughout study (for prospective cohort)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J. Matas, MD, Principal Investigator — University of Minnesota
Locations (7):
- United States (5):
  - University of Alabama - Division of Nephrology, Birmingham, Alabama
  - University of Iowa - Nephrology Division, Iowa City, Iowa
  - Hennepin County Medical Center - Division of Nephrology, Minneapolis, Minnesota
  - University of Minnesota Dept of Surgery - Transplantation Division, Minneapolis, Minnesota
  - Mayo Clinic - Division of Nephrology, Rochester, Minnesota
- Canada (2):
  - University of Alberta - Division of Nephrology & Immunology, Edmonton, Alberta
  - Health Sciences Center - Section of Nephrology, Winnipeg, Manitoba

REFERENCES:
- [Background] Hariharan S, Kasiske B, Matas A, Cohen A, Harmon W, Rabb H. Surrogate markers for long-term renal allograft survival. Am J Transplant. 2004 Jul;4(7):1179-83. doi: 10.1111/j.1600-6143.2004.00484.x. PMID 15196079
- [Background] Kasiske BL, Gaston RS, Gourishankar S, Halloran PF, Matas AJ, Jeffery J, Rush D. Long-term deterioration of kidney allograft function. Am J Transplant. 2005 Jun;5(6):1405-14. doi: 10.1111/j.1600-6143.2005.00853.x. PMID 15888048
- [Derived] Matas AJ, Helgeson E, Fieberg A, Leduc R, Gaston RS, Kasiske BL, Rush D, Hunsicker L, Cosio F, Grande JP, Cecka JM, Connett J, Mannon RB. Risk Prediction for Delayed Allograft Function: Analysis of the Deterioration of Kidney Allograft Function (DeKAF) Study Data. Transplantation. 2022 Feb 1;106(2):358-368. doi: 10.1097/TP.0000000000003718. PMID 33675321
- [Derived] Grande JP, Helgeson ES, Matas AJ. Correlation of Glomerular Size With Donor-Recipient Factors and With Response to Injury. Transplantation. 2021 Nov 1;105(11):2451-2460. doi: 10.1097/TP.0000000000003570. PMID 33273317
- [Derived] Oetting WS, Schladt DP, Dorr CR, Wu B, Guan W, Remmel RP, Ikle D, Mannon RB, Matas AJ, Israni AK, Jacobson PA; DeKAF Genomics and GEN03 Investigators. Analysis of 75 Candidate SNPs Associated With Acute Rejection in Kidney Transplant Recipients: Validation of rs2910164 in MicroRNA MIR146A. Transplantation. 2019 Aug;103(8):1591-1602. doi: 10.1097/TP.0000000000002659. PMID 30801535
- [Derived] Seibert SR, Schladt DP, Wu B, Guan W, Dorr C, Remmel RP, Matas AJ, Mannon RB, Israni AK, Oetting WS, Jacobson PA. Tacrolimus trough and dose intra-patient variability and CYP3A5 genotype: Effects on acute rejection and graft failure in European American and African American kidney transplant recipients. Clin Transplant. 2018 Dec;32(12):e13424. doi: 10.1111/ctr.13424. Epub 2018 Oct 31. PMID 30318646